CLINICAL TRIAL: NCT02702648
Title: Single-center, Double-blind, Randomized, Placebo-controlled, Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics (Including Food Effect), and Pharmacodynamics of an Oral Drug for Neurological Disorders in Healthy Subjects
Brief Title: First-in-man Study of Single and Multiple Ascending Doses of a New Drug for Neurological Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AC-082-101
Record Dates: First submitted 2016-02-24; First posted 2016-03-09 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Healthy Subjects
Keywords: healthy subjects; first-in-man; safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AC-082, Single Ascending Dose (Experimental): Subjects receive AC-082 at different single dose levels in a sequential manner, starting from 10 mg (number of cohorts and dose levels will depend on the safety and pharmacokinetic results of the previous cohort). Each subject can participate in only one dose level
  Interventions: Drug: AC-082
- Placebo, Single Ascending Dose (Placebo Comparator): Subjects receive a single dose of the matched placebo
  Interventions: Drug: Placebo
- AC-082, Multiple Ascending Dose (Experimental): Subjects receive AC-082 at different dose levels for 4 consecutive days in a sequential manner (dose levels and duration to be adapted according to the results of the single ascending dose cohorts). Each subject can participate in only one dose level
  Interventions: Drug: AC-082
- Placebo, Multiple Ascending Dose (Placebo Comparator): Subjects receive the matched placebo for 4 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AC-082 — Hard gelatin capsules for oral administration
  Arms: AC-082, Multiple Ascending Dose; AC-082, Single Ascending Dose
Drug: Placebo — Matched placebo capsules for oral administration
  Arms: Placebo, Multiple Ascending Dose; Placebo, Single Ascending Dose

SUMMARY:
The primary purpose of this first-in-man study is to investigate whether a new drug for neurological disorders is safe and well-tolerated when administered orally to healthy adults

ELIGIBILITY:
Key inclusion Criteria:

* Signed informed consent
* Healthy on the basis of physical examination,12-lead electrocardiogram and laboratory tests
* Males and females of non-childbearing potential, aged between 18 and 60 years (all inclusive)
* Women must have a negative serum pregnancy test at Screening and a negative urine pregnancy test predose on Day -1
* Body mass index (BMI) between 18.0 and 29.9 kg/m2 (inclusive)
* Systolic blood pressure (SBP), diastolic blood pressure (DBP) and pulse rate (PR) between 90-140 mmHg, 50-90 mmHg and 50-90 bpm (all inclusive), respectively

Key exclusion Criteria:

* History or clinical evidence of any disease and/or existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the study treatment
* Previous history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions
* Any circumstances or conditions, which, in the opinion of the Investigator, may affect full participation in the study or compliance with the protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2016-02-01; Primary Completion 2017-03-06 (Actual); Study Completion 2017-03-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to end of study (up to Day 11)
  Treatment-emergent adverse events and treatment-emergent serious adverse events
Changes from baseline in vital signs | Up to end of study (up to Day 11)
  Vital signs include diastolic and systolic blood pressure and pulse rate
Changes from baseline in ECG variables | Up to end of study (up to day 11)
  ECG variables are to be recorded at rest using a standard 12-lead ECG

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) following single ascending doses | From pre-dose on Day 1 to 96 hours post dose
  Cmax is derived from the observed plasma concentration-time curves
Time to reach Cmax (tmax) following single ascending doses | From pre-dose on Day 1 to 96 hours post dose
  tmax is derived from the observed plasma concentration-time curves
Terminal half-life [t(1/2)] following single ascending doses | From pre-dose on Day 1 to 96 hours post dose
Area under the plasma concentration-time curve (AUC) following single ascending doses | From pre-dose on Day 1 to 96 hours post dose
  AUC is defined for the time intervals from zero to time t of the last measured concentration above the limit of quantification [AUC(0-t)] and from zero to infinity [AUC(0-inf)]
Maximum plasma concentration (Cmax) following multiple ascending doses | Up to 96 hours following the last dose administration on Day 4
Time to reach Cmax (tmax) following multiple ascending doses | Up to 96 hours following the last dose administration on Day 4
Terminal half-life [t(1/2)] following multiple ascending doses | Up to 96 hours following the last dose administration on Day 4
  t(1/2) on the last day of dosing
Area under the plasma concentration-time curve during a dosing interval (AUCtau) | Day 1 and Day 4
  AUCtau is the area under the plasma concentration-time curve during a dosing interval

CONTACTS AND LOCATIONS:
Overall Officials: Karine Litherland, PhD, Study Director — Actelion
Locations (1):
- Investigator Site, Berlin, Germany